CLINICAL TRIAL: NCT02645227
Title: Platelet-rich Fibrin With 1.2% Rosuvastatin for the Treatment of Intrabony Defects in Chronic Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Platelet-rich Fibrin With 1.2% Rosuvastatin in Chronic Periodontitis Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and Head, Department of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/12/2013-14V
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Prolactin-Releasing Hormone; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Open flap debridement (OFD)
  Interventions: Procedure: Open flap debridement (OFD)
- Group 2 (Active Comparator): OFD with Platelet rich fibrin (PRF)
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)
- Group 3 (Active Comparator): OFD with PRF and 1.2% Rosuvastatin
  Interventions: Procedure: OFD with PRF and 1.2% Rosuvastatin

INTERVENTIONS:
Procedure: Open flap debridement (OFD) — Oral prophylaxis followed by OFD for treating bone defect
  Arms: Group 1
Procedure: OFD with Platelet rich fibrin (PRF) — Oral prophylaxis followed by OFD with PRF placement into the bone defect
  Arms: Group 2
Procedure: OFD with PRF and 1.2% Rosuvastatin — Oral prophylaxis followed by OFD with PRF and 1.2% Rosuvastatin placement into the bone defect
  Arms: Group 3

SUMMARY:
The present study is designed to evaluate the combined efficacy of Platelet Rich Fibrin (PRF) and 1.2% Rosuvastatin (RSV) with open flap debridement (OFD) in treatment of intrabony defects in chronic periodontitis patients

DETAILED DESCRIPTION:
ABSTRACT Background: Regenerative periodontal therapy encompasses the use of various bioactive agents that are not only inflammo-modulatory but also osteoclast-inhibitory or rather, osteostimulative. The hypolipidaemic Statin group of drugs, particularly Rosuvastatin (RSV), are known to be associated with alveolar bone formation and periodontal improvements. Platelet analogues like Platelet rich fibrin (PRF), being rich sources of growth factors, have also come into widespread periodontal regenerative use. The aim of the study is to evaluate and compare the efficacy of open-ﬂap debridement (OFD) with or without PRF or PRF + 1.2% RSV gel in the treatment of intrabony defects (IBDs) in chronic periodontitis (CP) patients.

Methods: Ninety individuals with a total of 90 IBDs were randomly assigned to one of the 3 treatment groups: 1) OFD alone, 2) OFD + PRF and 3) OFD + PRF + 1.2% RSV gel placement. Plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), clinical attachment (CA) level and IBD depth were recorded at baseline and at 9 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy with CP diagnosis16 having probing depth (PD) ≥5mm, clinical attachment (CA) level ≥3mm and vertical bone loss ≥3mm on intraoral periapical radiographs (IOPAR) without any antibiotic or periodontal therapy in the last 6 months.

Exclusion Criteria:

* History of statin allergy, statin therapy, any systemic condition or medication altering the periodontal condition, immune-compromised state, hematologic disorders, insufﬁcient platelet count (<200,000/mm3), aggressive periodontitis, substance/tobacco abuse and lactating and pregnant females.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
defect depth reduction (%) | Change from baseline to 9 months
  assessed in percentage

SECONDARY OUTCOMES:
probing depth (mm) | Change from baseline to 9 months
  measured in mm
clinical attachment level (mm) | Change from baseline to 9 months
  measured in mm
modified sulcus bleeding index | Change from baseline to 9 months
  scale from 0-3
plaque index | Change from baseline to 9 months
  scale from 0-3

CONTACTS AND LOCATIONS:
Overall Officials: Avani Pradeep, MDS, Study Director — Government Dental Colleege & Research Institute, Bangalore
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India